CLINICAL TRIAL: NCT04104347
Title: Does Metacognitive Training Improve Insight and Clinical Outcomes in Schizophrenia?
Brief Title: Metacognitive Training and Insight in Schizophrenia
Acronym: MCT-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Universidad Autonoma de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC044-19_FJD-HRJC
Record Dates: First submitted 2019-07-31; First posted 2019-09-26 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: schizophrenia spectrum disorders; metacognitive training; insight; ecological momentary assessment
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Self-Help Groups

STUDY DESIGN:
Intervention Model Description: This single-center, assessor-blind, parallel-group, randomised clinical trial (RCT) aims to investigate the efficacy of MCT for improving insight (primary outcome), including clinical and cognitive insight, which will be measured by the Schedule for Assessment of Insight (Expanded version) (SAI-E) and the Beck Cognitive Insight Scale (BCIS), respectively, in (at least) n=126 outpatients with SSD at three points in time: i) at baseline (Time 0); ii) after treatment (Time 1) and iii) at 1-year follow-up (Time 2). SSD patients receiving MCT and controls attending a non-intervention support group will be compared on insight level changes and several clinical and cognitive secondary outcomes at Time 1 and at Time T2, whilst adjusting for baseline data. Ecological momentary assessment (EMA) will be piloted to assess functioning in a subsample of participants.
Who Masked: Outcomes Assessor
Masking Description: After the baseline (Time 0) assessment participants are randomised to either MCT or the control group through a computerized plan (no stratification factors) in blocks of 10 subjects (maximum number of each group) and assessor-patient blind. Only one co-principal investigator of the project (EBG) has access to the randomisation plan, but the assessor (JDLM) is not informed of the patient's allocation arm. Also, big efforts will be made on the ground to reduce the risk that the assessor (JDLM) may become accidentally unblinded and patients are reminded that they should not disclose their group assignment at any time. At the end of the baseline assessment, participants receive an envelope with the intervention assignment from an independent administrator who is not involved in the research team. Hence, assessor-blindness is guaranteed at all times throughout the study period since the assessor (JDLM) is not involved in the randomization plan or the active interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metacognitive training (MCT) (Experimental)
  Interventions: Other: Metacognitive training (MCT)
- Support group (Active Comparator)
  Interventions: Other: Support group

INTERVENTIONS:
Other: Metacognitive training (MCT) — Metacognitive Training (MCT) was first developed in Germany in 2007 by Steffen Moritz and Todd Woodward (Moritz & Woodward, 2007) targeting positive psychotic symptoms of patients with schizophrenia. MCT aims to change cognitive biases leading to delusional beliefs and consists of ten group sessions focused on different topics (Modules) as follows: Attributional Style (Module 1), Jumping to Conclusions (Modules 2 and 7), Changing Beliefs (Module 3), Empathy (Modules 4 and 6), Memory (Modules 5), Depression and Self-Esteem (Module 8) and two additional modules, namely Self-Esteem (Module 9) and Stigma (Module 10). Modules 8 (Self-Esteem), 9 (Self-Esteem) and 10 (Stigma) can be delivered together as one session so the intervention totals eight weekly group (3-10 participants) sessions. The MCT manual is available at: http://www.uke.de/mkt and was directly supervised by Steffen Moritz.
  Arms: Metacognitive training (MCT)
Other: Support group — Controls will attend eight weekly support groups. Seven group sessions will focus on the following topics: 1) basic activities of daily living (BADL), 2) instrumental activities of daily living (IADL), 3) physical health, 4) press-based work, 5) psychoeducation on emotions, 6) psychoeducation on illness, 7) social and family relationships. One additional session will give participants some time to openly raise general issues and concerns which were not discussed during the above sessions. Controls will be encouraged to attend these group sessions from which they are likely to benefit. While not an intervention as such, this should turn into enough incentive to reach similar attendance rates in both arms of the RCT.
  Arms: Support group

SUMMARY:
Although insight in schizophrenia spectrum disorders (SSD) has been associated with positive outcomes, the effect size of previous treatments on insight has been relatively small to date. The metacognitive basis of insight suggests that metacognitive training (MCT) may improve insight and clinical outcomes in SSD, although this remains to be established.

This single-center, assessor-blind, parallel-group, randomised clinical trial (RCT) aims to investigate the efficacy of MCT for improving insight (primary outcome), including clinical and cognitive insight, which will be measured by the Schedule for Assessment of Insight (Expanded version) (SAI-E) and the Beck Cognitive Insight Scale (BCIS), respectively, in (at least) n=126 outpatients with SSD at three points in time: i) at baseline (Time 0); ii) after treatment (Time 1) and iii) at 1-year follow-up (Time 2). SSD patients receiving MCT and controls attending a non-intervention support group will be compared on insight level changes and several clinical and cognitive secondary outcomes after treatment and at follow-up, whilst adjusting for baseline data. Ecological momentary assessment (EMA) will be piloted to assess functioning in a subsample of participants.

This will be the first RCT testing the effect of group MCT on multiple insight dimensions (as primary outcome) in a sample of unselected patients with SSD, including several secondary clinically relevant outcomes, namely symptom severity, functioning, which will also be evaluated with EMA, hospitalizations and suicidal behaviour.

DETAILED DESCRIPTION:
INTRODUCTION:

Schizophrenia and related disorders remain associated with relatively poor psychosocial outcomes. Impaired insight has been reported to be the strongest predictor of this poor outcome in psychotic disorders. However, the effect size of previous treatments on insight changes in psychotic disorders has been relatively small to date, which may have been the result of not tackling the actual underpinnings of insight in psychosis.

Several theories have been proposed to explain what underlies 'lack of insight' in schizophrenia spectrum disorders. First, lack of insight could be viewed as having a function in terms of being protective or preserving self-esteem, i.e., a denial mechanism. Second, lack of insight may also be considered as a primary symptom of the disorder. Third, the neurocognitive basis of insight was in part supported by a meta-analysis, which also suggested that other variables, namely metacognition, which was defined as 'the ability to think of one's and others' thinking', may affect insight. Indeed, patients with schizophrenia have been reported to show metacognitive deficits and poorer metacognitive performance is linked with impaired insight in schizophrenia. Metacognitive training (MCT) may therefore improve insight, which should also have a positive impact on clinical outcomes, although no previous randomized clinical trials (RCT) have investigated this.

MCT was first developed by Steffen Moritz and Todd Woodward and is available at no cost at: http://www.uke.de./mct. Since then, one systematic review and four meta-analyses have replicated the positive effects of MCT on positive symptoms, particularly delusions, when compared with 'treatment as usual' (TAU), although one meta-analysis failed to show such an association. However, to the best of our knowledge no definitive randomised clinical trial (RCT) using MCT has considered insight as primary outcome to date, although three previous RCTs found other non-MCT metacognitively oriented therapies to improve insight in first-episode psychosis and schizophrenia.

Clinical and cognitive insight are different, albeit related, concepts. There has been a growing interest in clinical insight in psychosis since the multidimensional model of insight proposed by David, which encompasses three different, albeit overlapping, dimensions - illness recognition, symptom relabelling and treatment compliance - and has been consistently replicated ever since. Multidimensional measurement scales, such as the Scale of Uawareness of Mental Disorder (SUMD) and the Schedule for Assessment of Insight (SAI-E), were also devised for research. Cognitive insight is a core metacognitive domain which refers to the person's ability to evaluate and correct his/her own distorted beliefs and misinterpretations (self-reflectiveness) and the tendency to overconfidence in one's conclusions (self-certainty).

The main aim of this RCT is to test whether MCT can improve insight, including clinical and cognitive insight, in patients with schizophrenia over a 1-year follow-up. As secondary aims, the effect of MCT-related insight changes on clinical outcomes, including symptomatic severity, hospitalizations, suicidal behaviour and psychosocial Functioning, will be investigated. In addition, the investigators will pilot the use of ecological momentary assessment (EMA) via two web-based applications - www.MEmind.net and the Evidence-Based Behaviour platform eB2 app - to measure functioning in a subsample of participants.

Specifically, the following five hypotheses are to be tested: i) that MCT will result in higher cognitive and clinical insight levels and that MCT-induced insight improvement will be linked with (compared with controls): ii) reduced symptom severity and iii) lower risk of hospitalizations, iv) lower suicide rates and v) better functioning.

METHODS:

Study design This is a single-center, assessor-blind, parallel group, two-armed randomised controlled trial (RCT) over a 1-year follow-up period. Participants will be assessed at baseline, following which they will be randomised to either group MCT (experimental group) or a support group (control group) and they will be reassessed after treatment, i.e., at approximately 8 weeks, and at 1-year follow-up.

The study protocol has been approved by the local Research Ethics Committee of the Instituto de Investigación Sanitaria (IIS)-Fundación Jiménez Díaz (Madrid, Spain), from which patients will be recruited as detailed below, and registered as RCT-EC044-19_FJD_HRJC.

Recruitment process:

Recruitment will occur at the outpatient clinic known as Centro de Salud Mental de Arganzuela, which is part of Instituto Fundacion Jimenez Diaz, that is, the 'sponsor', at which two consultant psychiatrists and one consultant psychologist will refer potential candidates to the principal investigator of the project (JDLM) to arrange a first pre-recruitment interview during which the relevant information of the project is explained to the candidate in lay terms, including an information leaflet. Those agreeing to participate in the study are screened against the above inclusion/exclusion criteria at this point. Those who are found to fulfill the study selection criteria undertake a neurocognitive assessment. Specifically, the WAIS-IV is administered by a MSc-level clinical psychologist in order to rule out an IQ≤70, which is an exclusion criterion. Those with an IQ>70 are administered the Trail Making Test (TMT), which assesses executive function and has been found to correlate with insight scores in psychosis patients, shortly after the WAIS-IV in order to complete the baseline neurocognitive assessment at this point.

After a short break of around 5 minutes, the 'assessor' (JDLM) performs the MINI International Psychiatric Interview to confirm the diagnosis of psychosis and conducts the psychopathological, insight, metacognitive and functioning assessments detailed below. Also, a set of demographic and clinical variables, which are listed below, are collected at this baseline interview.

All participants will be encouraged to continue taking medication as prescribed by the treating consultant psychiatrist, usually antipsychotics, and to receive non-metacognitive oriented psychotherapy, such as psychoeducation. There will be no restrictions on medication changes over the trial, which can be made by the treating consultant at any time, although medication-related variables will be considered in secondary analyses as potential mediators/confounders. Participants are informed of their right to drop out of the study at any time without having to disclose a specific reason, which will have no implications on treatment or service provision. Participants are not compensated with any amount of money for completing the assessments and/or receiving the interventions, namely MCT or attending a weekly support group.

Randomisation and assessor-blindness:

After the baseline (Time 0) assessment participants are randomised to either MCT or the support group, both of which are run by two researchers, through a computerized plan (no stratification factors) in blocks of 10 subjects (maximum number of each group) and assessor (JDLM)-patient blind. Only one co-principal investigator of the project (EBG) has access to the randomisation plan, but the assessor (JDLM) is not informed of the patient's allocation group, thus ensuring assessor-blindness. Since the patient may find out what intervention he/she is receiving the study cannot be considered to be 'double-blind', although it is 'single-blind', that is, 'assessor-blind'. Also, big efforts will be made on the ground to reduce the risk that the assessor (JDLM) may become accidentally unblinded and patients are reminded that they should not disclose their group assignment at any time. At the end of the baseline assessment, participants receive an envelope with the intervention assignment from an independent administrator who is not involved in the research team. A reminder mobile text-message is also sent to participants within the next 24 hours with the group details (date, time and venue), which is also re-sent again during the 24 hours prior to the appointment, which is very similar to our routine clinical practice. Hence, assessor-blindness is guaranteed at all times throughout the study period since the assessor (JDLM) is not involved in the randomization plan or the active interventions.

Assessments:

Participants will be assessed at three timepoints: i) at baseline (Time 0); ii) after treatment (Time 1); iii) at 1-year follow-up (Time 2). Data on different variables will be collected at each of these assessments.

The assessor (JDLM) completed a rater-training workshop and received individual training in which they were observed as they assessed pilot patients by using the project scales explained below under the supervision of a senior consultant psychiatrist with expertise in the use of these instruments (EBG).

Additional variables:

Demographic and clinical data:

At baseline data on the following demographic and clinical variables will be collected: gender, age at the study inception, nationality, ethnicity, marital status, education level, living status, employment status, ICD-10 diagnosis, duration of untreated psychosis, number of previous admissions, number, date and method of previous suicidal acts, current medications, alcohol/illicit drugs dependence (present/absent), medical comorbidities (present/absent) family history of mental illness (present/absent).

Marital status, living status and employment status will be reassessed at 1-year follow-up as measures of functioning.

Premorbid adjustment:

Premorbid adjustment, which can be defined as 'the degree of achievement of developmental goals' will be retrospectively rated with the Premorbid Adjustment Scale (PAS). Specifically, the PAS provides scores on the level of adjustment over i) childhood (to age 11), ii) early adolescence (age 11-15), iii) late adolescence (age 15-17) and iv) adulthood (age ≥18). With regard to childhood and adolescence, items inquiry about sociability and social withdrawal, peer relationships, scholastic performance, adaptation to school and ability to form socio-sexual relationships. The questions regarding adulthood focus on social relationships by asking about educational achievement, social relationships and level of interest in, and enjoyment of, major life activities, such as work or family.

Neurocognition:

The neurocognitive assessment battery, which will be administered at the three assessments, will include the short version of the Wechsler Adult Intelligence Scale (WAIS) Revised, which estimates current intelligence quotient (IQ), and the Trail Making Test (TMT), which assesses executive function. Subtracting time in seconds to complete TMT task B minus time in seconds to complete TMT task A gives a measure of executive function, whilst controlling for processing speed.

Metacognition:

Three metacognitive tasks will be completed by participants at baseline, after treatment and at 1-year follow-up:

* Jumping to Conclusions (JTC) will be determined with the beads task. During this task, the individual is asked to decide the jar to which the extracted bead belongs on the basis of probability (in task 1 the probability is 85:15, while in task 2 the probability is 60:40). 'JTC' is considered as making a decision after extracting one or two beads.
* The Hinting Task will be used to measure Theory of Mind (ToM) performance. Learning is avoided by using different stories at the three assessments. Cronbach's α was good (0.64) for the Spanish version.
* In addition, the Emotional Recognition Test Faces, which is composed of 20 different pictures representing people's emotions, will be used to evaluate ToM.

Statistical analysis:

Participants' data will be analysed at the end of the study on an intention-to-treat (ITT) basis, thus including all patients with baseline information available. Imputation methods will be used to estimate missing values. All the analyses will be performed with the Statistical Package for Social Science version 25.0 (SPSS Inc., Chicago, IL, USA).

First, demographic and clinical characteristics of groups (MCT and controls), including insight measures, will be compared at baseline so parametric and non-parametric tests will be used as appropriate. Also, for descriptive purposes, between-arm completion rates differences will be analysed at the end of the study.

Second, in order to investigate the primary outcome of the study, namely insight changes over the trial period, univariate analysis of covariance (ANCOVA) models will examine between-group differences (MCT and controls) in the SAI-E and BCIS total and subtotal scores changes from Time 0 to Time 1 and from Time 0 to Time 2 (as the dependent variable), whilst adjusting for baseline data. Hence, the effects of treatment (independent of time) and treatment group allocation*time interactions on insight changes will be investigated. The investigators will also explore within-group scores changes between Time 0, Time 1 and Time 2. Specifically, effect sizes (Cohen's d) and the corresponding 95% confidence intervals (CI) will be estimated from the imputed datasets for between- and within-group insight scores changes. In accordance with Cohen's conventions, effect sizes will be classified as 'small' (d<0.2), 'medium' (d=0.2-0.5) or 'large' (d>0.8). Due to multiple testing and the subsequent risk of type I error, results will be adjusted using Bonferroni correction.

Third, for the secondary outcomes evaluated with continuous variables, i.e., symptom severity (PANSS and CDSS) and functioning (GAF, SDLS and WHODAS), analogous ANCOVA models will be used. For those binary secondary outcomes, namely suicidal behaviour and readmissions, survival analyses, i.e., multivariable Cox regression models, will model time to the outcome event (i.e., first suicidal event or hospital admission, respectively) or the censoring date as appropriate, whilst adjusting for baseline variables.

Finally, variables inter-relationships over the trial period will be examined by means of path analysis through structural equation modeling, thus testing the effect of putative mediators/moderators/confounders/covariates, including neurocognition measures, on the above associations.

Power calculations and estimation of sample size:

Given that the mean SAI-E score for psychosis patients is 13/28 with a standard deviation of around 6, a difference of 2 points (e.g., 13 vs. 15) between groups (e.g., MCT vs. controls), which is considered to be clinically meaningful, is equivalent to an effect size of 0.33 with a two-tailed alpha significant level set at 5%. Under these assumptions, for reaching a sufficient statistical power of β=80% at the end of the study, n=63 subjects in each arm will be needed, that is, a total sample size of N=126 patients, who will be analysed at the end of the study on an intention-to-treat (ITT) basis. Attrition rates in previous RCTs investigating MCT effects on symptoms were low (approximately 10%). However, since participants will be followed-up over a more prolonged period (1 year) the investigators have conservatively assumed a much higher drop-out rate of 50%. Under this assumption, the study will be carried out with an initial sample size of N=252 patients, i.e., n=126 participants in each group/arm at the study inception, which will also allow both ITT and 'per protocol' analyses with sufficient power.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-64 years, both inclusive
* Diagnosis: schizophrenia spectrum disorder (F20-F29, ICD-10)
* Outpatient status

Exclusion Criteria:

* IQ≤70 as measured by the short form of the Wechsler Adults Intelligence Scale (WAIS) (Wechsler, 1981).
* History of head injury and/or a neurological condition.
* Having received a metacognitively oriented therapy within the previous 12 months.
* Low level of Spanish.
* Lack of cooperativeness with the assessment and/or "intervention".

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive insight | Change in cognitive insight will be evaluated after treatment at 2 months (Month 2) and at 12 months (Month 12). Changes from baseline (Day 0) score to Month 2 (Month 2 - Day 0) and from baseline to Month 12 (Month 12 - Day 0) will be calculated.
  The Spanish version of the Beck Cognitive Insight Scale (BCIS), which is a 15-item self-administered scale which evaluates self-reflectiveness (9 items) and self-certainty (6 items). Each item is rated within a Likert scale ranging from 0 ("I disagree") to 4 ("I totally agree") so they can be summed up to create two subtotal scores, namely self-reflectiveness (ranging from 0 to 36, i.e., higher scores, better insight) and self-certainty (ranging from 0 to 24, where higher scores indicate worse insight). A composite index (CI) can also be calculated by subtracting self-certainty from self-reflectiveness so CI higher scores indicate better insight. Internal consistency was found to be acceptable (Cronbach's α=0.60-0.68).
Change in clinical insight | Change in clinical insight will be assessed after-treatment at 2 months (Month 2) and at 12 months or follow-up (Month 12). Changes from baseline (Day 0) scores to Month 2 (Month 2-Day0) and from baseline to 12 months (Month 12-Day 0) will be calculated.
  The Spanish version of the Schedule for Assessment of Insight (expanded version) (SAI-E) will assess clinical insight. The SAI-E takes the form of a semi-structured interview which enquires about different aspects of insight by means of items ranging from 0 to 3, 4 ,5, or 7. The SAI-E provides scores on three insight dimensions in line with David's model - illness recognition (scores ranging from 0 to 10), symptom relabeling (scores ranging from 0 to 12), treatment compliance (range: 0-6) - and a total insight score (ranging from 0 to 28). Higher scores indicate better insight.

SECONDARY OUTCOMES:
Change in psychotic symptoms severity | Change in psychotic symptoms severity will be assessed at 2 months (Month 2) and at 12 months (Month 12). Changes from baseline (Day 0) scores to 2 months (Month 2 - Day 0) and from baseline to 12 months (Month 12 - Day 0) will be calculated.
  The Spanish version of the Positive and Negative Syndrome Scale (PANSS) will be used to measure psychotic symptoms severity. The PANSS includes 30 items, each of which is rated within a Likert scale, with scores ranging from 1(absent) to 7 (most severe). The PANSS includes 7 items enquiring about positive symptoms (so this subscale score ranges from 7 to 49), 7 ítems on negative symptoms (this subscale score ranges from 7 to 49) and 16 items about general psychopathology (this subscale score ranges from 16 to 112). They can be therefore summed up to create a total score, which ranges from 30 to 210, where higher scores indicate more severe psychotic symptoms.
Change in depressive symptoms severity | Change in depressive symptoms severity will be assessed at 2 months (Month 2) and at 12 months (Month 12). Changes from baseline (Day 0) scores to 2 months (Month 2 - Day 0) and from baseline to 12 months (Month 12 - Day 0) will be calculated.
  The Calgary Depression Scale for Schizophrenia (CDSS). The CDSS is formed of 9 items enquiring about symptoms of depression over the last two weeks. Each item is rated within a Likert Scale from 0 (absent) to 3 (most severe), which can be summed up to create a total score which therefore ranges from 0 to 27 (higher scores indicate more severe depressive symptoms).
Hospitalizations | Number of hospitalizations and length of stay will be considered over the 1-year follow-up trial period.
  Number of hospitalizations, i.e., time to hospitalization (i.e., survival analyses, see statistical analyses below), and total number of days in hospital will be considered. Mental health presentations to the emergency department will be included in secondary analyses.
Time to first suicidal event | Data on suicidal behaviour will be collected at 12-month follow-up, which is the trial period.
  Time to first suicidal event, including suicide attempts and suicide completions, whichever came sooner, will be analysed by means of survival analyses in relation to baseline data at the end for the trial.
Change in General Functioning | Change in general functioning will be determined at 2 months (Month 2) and at 12 months (Month 12). Changes in scores from baseline (Day 0) to 2 months (MOnth 2 - Day 0) and from baseline to 12 months (Month 12 - Day 0) will be calculated.
  General Functioning will be recorded through the Global Assessment of Functioning (GAF), which is a rater-based scale widely used by mental health professionals to rate the social, occupational and psychological level of functioning of the patient. Scores range from 0 to 100, where higher scores indicate better functioning.
Change in disability | Change in disability will be assessed at 2 months (Month 2) and at 12 months (Month 12). Changes in scores from baseline (Day 0) to 2 months (Month 2 - Day 0) and from baseline to 12 months (Month 12 - Day 0) will be calculated.
  The World Health Organization Disability Schedule (WHODAS) will be used to evaluate participants' disablity. The WHODAS includes 12 questions enquiring about the level of difficulty to carry out day-to-day activities as rated by the individual. Each item is rated within a Likert scale, with scores ranging from 0 (no difficulty) to 4 (highest level of difficulty). The items scores can be summed up to create total scores which range from 0 to 48, where higher scores indicate greater disability.
Change in quality of life | Change in quality of life will be determined at 2 months (Month 2) and at 12 months (Month 12). Changes in scores from baseline (Day 0) to 2 months (Month 2 - Day 0) and from baseline to 12 months (Month 12 - Day 0) will be calculated.
  Quality of life will be measured by the Spanish version of the Satisfaction Life Domains Scale (SLDS), which assesses satisfaction with the patient's life as a whole. The SLDS is a self-rated 15-item scale, each of which enquiries about different domains such as health or finances and ranges from 1 (very dissatisfied) to 7 (very satisfied). Total scores therefore range from 15 to 105, with higher scores indicating better quality of life.
Ecological momentary assessment | Memind and eB2 will continuously collect patient's data on behaviour and functioning in real time throughout the trial period from the day of the baseline assessment (Day 0) to the end of the 12-month follow-up period (Month 12).
  Two web-based applications installed in participants' smartphones, namely Memind (www.memind.net) and eB2, will record data on sociodemographic, social, occupational, behavioural, mobility and location variables with- (memind) and without (eB2) participant's collaboration.

CONTACTS AND LOCATIONS:
Overall Officials: Javier-David Lopez-Morinigo, MB BS, PhD, Principal Investigator — Hospital Universitario Fundacion Jiménez Díaz. Universidad Autónoma de Madrid. Madrid (Spain)
Locations (1):
- Hospital Universitario Fundación JIménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to other researchers, provided the dataset access rules detailed below are complied with.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the end of the baseline data collection, that is, by April 2020, baseline data will become available to other researchers, provided the access criteria below are complied with.
Access Criteria: * An application needs to be made by an independent researcher which will have to specify:
  * Variables on which data are requested need to be listed.
  * Inclusion/exclusion criteria of participants.
  * Brief summary of the study protocol (e.g. specific outcome measures).
  * Statistical analysis plan
  * Results publication plan. Prior to submitting a manuscript for publication including findings from our dataset, this manuscript will have to be approved, including the relevant email, by the principal investigator of this project, (JDLM).
  * Ethical approval from the applicant's local Research Ethics Committee.
  * Ethical approval from our local Research Ethics Committee.

REFERENCES:
- [Background] Morgan C, Lappin J, Heslin M, Donoghue K, Lomas B, Reininghaus U, Onyejiaka A, Croudace T, Jones PB, Murray RM, Fearon P, Doody GA, Dazzan P. Reappraising the long-term course and outcome of psychotic disorders: the AESOP-10 study. Psychol Med. 2014 Oct;44(13):2713-26. doi: 10.1017/S0033291714000282. Epub 2014 Feb 26. PMID 25066181
- [Background] Lysaker PH, Pattison ML, Leonhardt BL, Phelps S, Vohs JL. Insight in schizophrenia spectrum disorders: relationship with behavior, mood and perceived quality of life, underlying causes and emerging treatments. World Psychiatry. 2018 Feb;17(1):12-23. doi: 10.1002/wps.20508. PMID 29352540
- [Background] Pijnenborg GH, van Donkersgoed RJ, David AS, Aleman A. Changes in insight during treatment for psychotic disorders: a meta-analysis. Schizophr Res. 2013 Mar;144(1-3):109-17. doi: 10.1016/j.schres.2012.11.018. Epub 2013 Jan 8. PMID 23305612
- [Background] Pijnenborg GH, Timmerman ME, Derks EM, Fleischhacker WW, Kahn RS, Aleman A. Differential effects of antipsychotic drugs on insight in first episode schizophrenia: Data from the European First-Episode Schizophrenia Trial (EUFEST). Eur Neuropsychopharmacol. 2015 Jun;25(6):808-16. doi: 10.1016/j.euroneuro.2015.02.012. Epub 2015 Apr 20. PMID 25907250
- [Background] Cooke MA, Peters ER, Kuipers E, Kumari V. Disease, deficit or denial? Models of poor insight in psychosis. Acta Psychiatr Scand. 2005 Jul;112(1):4-17. doi: 10.1111/j.1600-0447.2005.00537.x. PMID 15952940
- [Background] Cuesta MJ, Peralta V, Campos MS, Garcia-Jalon E. Can insight be predicted in first-episode psychosis patients? A longitudinal and hierarchical analysis of predictors in a drug-naive sample. Schizophr Res. 2011 Aug;130(1-3):148-56. doi: 10.1016/j.schres.2011.04.032. Epub 2011 May 31. PMID 21632216
- [Background] Aleman A, Agrawal N, Morgan KD, David AS. Insight in psychosis and neuropsychological function: meta-analysis. Br J Psychiatry. 2006 Sep;189:204-12. doi: 10.1192/bjp.189.3.204. PMID 16946354
- [Background] Flavell JH. Metacognition and cognitive monitoring: a new area of cognitive-developmental inquiry. Am Psychol. 1979;34:906-911
- [Background] Wells A, Purdon C. Metacognition and cognitive-behaviour therapy: A special issue. Clin Psychol Psychoter. 1999;6(2):71-2.
- [Background] Beck AT, Baruch E, Balter JM, Steer RA, Warman DM. A new instrument for measuring insight: the Beck Cognitive Insight Scale. Schizophr Res. 2004 Jun 1;68(2-3):319-29. doi: 10.1016/S0920-9964(03)00189-0. PMID 15099613
- [Background] Dimaggio G, Lysaker, PH. Metacognition and Severe Adult Mental Disorders. From Research to Treatment. 1st ed. New York; Routledge; 2010.
- [Background] Nair A, Palmer EC, Aleman A, David AS. Relationship between cognition, clinical and cognitive insight in psychotic disorders: a review and meta-analysis. Schizophr Res. 2014 Jan;152(1):191-200. doi: 10.1016/j.schres.2013.11.033. Epub 2013 Dec 16. PMID 24355529
- [Background] Moritz S, Woodward T S. Metacognitive Training for schizophrenia patients (MCT): A pilot study on feasibility, treatment adherence, and subjective efficacy. German Journal of Psychiatry. 2007;10(3):69-78.
- [Background] Moritz S, Andreou C, Schneider BC, Wittekind CE, Menon M, Balzan RP, Woodward TS. Sowing the seeds of doubt: a narrative review on metacognitive training in schizophrenia. Clin Psychol Rev. 2014 Jun;34(4):358-66. doi: 10.1016/j.cpr.2014.04.004. Epub 2014 May 6. PMID 24866025
- [Background] Jiang J, Zhang L, Zhu Z, Li W, Li C. Metacognitive training for schizophrenia: a systematic review. Shanghai Arch Psychiatry. 2015 Jun 25;27(3):149-57. doi: 10.11919/j.issn.1002-0829.215065. PMID 26300597
- [Background] Eichner C, Berna F. Acceptance and Efficacy of Metacognitive Training (MCT) on Positive Symptoms and Delusions in Patients With Schizophrenia: A Meta-analysis Taking Into Account Important Moderators. Schizophr Bull. 2016 Jul;42(4):952-62. doi: 10.1093/schbul/sbv225. Epub 2016 Jan 8. PMID 26748396
- [Background] Liu YC, Tang CC, Hung TT, Tsai PC, Lin MF. The Efficacy of Metacognitive Training for Delusions in Patients With Schizophrenia: A Meta-Analysis of Randomized Controlled Trials Informs Evidence-Based Practice. Worldviews Evid Based Nurs. 2018 Apr;15(2):130-139. doi: 10.1111/wvn.12282. Epub 2018 Feb 28. PMID 29489070
- [Background] Philipp R, Kriston L, Lanio J, Kuhne F, Harter M, Moritz S, Meister R. Effectiveness of metacognitive interventions for mental disorders in adults-A systematic review and meta-analysis (METACOG). Clin Psychol Psychother. 2019 Mar;26(2):227-240. doi: 10.1002/cpp.2345. Epub 2018 Dec 16. PMID 30456821
- [Background] van Oosterhout B, Smit F, Krabbendam L, Castelein S, Staring AB, van der Gaag M. Metacognitive training for schizophrenia spectrum patients: a meta-analysis on outcome studies. Psychol Med. 2016 Jan;46(1):47-57. doi: 10.1017/S0033291715001105. Epub 2015 Jul 20. PMID 26190517
- [Background] Vohs JL, Leonhardt BL, James AV, Francis MM, Breier A, Mehdiyoun N, Visco AC, Lysaker PH. Metacognitive Reflection and Insight Therapy for Early Psychosis: A preliminary study of a novel integrative psychotherapy. Schizophr Res. 2018 May;195:428-433. doi: 10.1016/j.schres.2017.10.041. Epub 2017 Nov 3. PMID 29108671
- [Background] de Jong S, van Donkersgoed RJM, Timmerman ME, Aan Het Rot M, Wunderink L, Arends J, van Der Gaag M, Aleman A, Lysaker PH, Pijnenborg GHM. Metacognitive reflection and insight therapy (MERIT) for patients with schizophrenia. Psychol Med. 2019 Jan;49(2):303-313. doi: 10.1017/S0033291718000855. Epub 2018 Apr 25. PMID 29692285
- [Background] Pijnenborg GHM, de Vos AE, Timmerman ME, Van der Gaag M, Sportel BE, Arends J, Koopmans EM, Van der Meer L, Aleman A. Social cognitive group treatment for impaired insight in psychosis: A multicenter randomized controlled trial. Schizophr Res. 2019 Apr;206:362-369. doi: 10.1016/j.schres.2018.10.018. Epub 2018 Nov 12. PMID 30429078
- [Background] David AS. Insight and psychosis. Br J Psychiatry. 1990 Jun;156:798-808. doi: 10.1192/bjp.156.6.798. PMID 2207510
- [Background] Amador XF, David AS. Insight and Psychosis. Awareness of Illness in Schizophrenia and Related Disorders. 2nd ed. New York: Oxford University Press; 2004.
- [Background] Amador XF, Strauss DH, Yale SA, Flaum MM, Endicott J, Gorman JM. Assessment of insight in psychosis. Am J Psychiatry. 1993 Jun;150(6):873-9. doi: 10.1176/ajp.150.6.873. PMID 8494061
- [Background] . Kemp R, David AS. Insight and Compliance. In: Blackwell, B editor. Treatment Compliance and the Therapeutic Alliance in Serious Mental Illness. The Netherlands: Harwood Academic Publishers; 1997. p. 61-86
- [Background] Barrigon ML, Berrouiguet S, Carballo JJ, Bonal-Gimenez C, Fernandez-Navarro P, Pfang B, Delgado-Gomez D, Courtet P, Aroca F, Lopez-Castroman J, Artes-Rodriguez A, Baca-Garcia E; MEmind study group. User profiles of an electronic mental health tool for ecological momentary assessment: MEmind. Int J Methods Psychiatr Res. 2017 Mar;26(1):e1554. doi: 10.1002/mpr.1554. Epub 2017 Mar 9. PMID 28276176
- [Background] Berrouiguet S, Ramirez D, Barrigon ML, Moreno-Munoz P, Carmona Camacho R, Baca-Garcia E, Artes-Rodriguez A. Combining Continuous Smartphone Native Sensors Data Capture and Unsupervised Data Mining Techniques for Behavioral Changes Detection: A Case Series of the Evidence-Based Behavior (eB2) Study. JMIR Mhealth Uhealth. 2018 Dec 10;6(12):e197. doi: 10.2196/mhealth.9472. PMID 30530465
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Wechsler D. The Wechsler Adult Intelligence Scale-Revised. New York: The Psychological Corporation; 1981.
- [Background] Reitan R. Validity of the Trail Making Test as an indicator of organic brain damage. Perceptual and Motor Skills. 1958;8(3):271-6
- [Background] Lopez-Morinigo JD, Di Forti M, Ajnakina O, Wiffen BD, Morgan K, Doody GA, Jones PB, Ayesa-Arriola R, Canal-Rivero M, Crespo-Facorro B, Murray RM, Dazzan P, Morgan C, Dutta R, David AS. Insight and risk of suicidal behaviour in two first-episode psychosis cohorts: Effects of previous suicide attempts and depression. Schizophr Res. 2019 Feb;204:80-89. doi: 10.1016/j.schres.2018.09.016. Epub 2018 Sep 22. PMID 30253893
- [Background] Soriano-Barceló J, López-Moríñigo JD, Ramos-Ríos R, Rodríguez-Zanabria EA, David AS. Insight assessment in psychosis and psychopathological correlates: Validation of the Spanish version of the Schedule for Assessment of Insight - Expanded Version. Eur J Psychiat. 2016;30(1):55-65
- [Background] Sanz M, Constable G, Lopez-Ibor I, Kemp R, David AS. A comparative study of insight scales and their relationship to psychopathological and clinical variables. Psychol Med. 1998 Mar;28(2):437-46. doi: 10.1017/s0033291797006296. PMID 9572100
- [Background] Morgan KD, Dazzan P, Morgan C, Lappin J, Hutchinson G, Suckling J, Fearon P, Jones PB, Leff J, Murray RM, David AS. Insight, grey matter and cognitive function in first-onset psychosis. Br J Psychiatry. 2010 Aug;197(2):141-8. doi: 10.1192/bjp.bp.109.070888. PMID 20679268
- [Background] Gutierrez-Zotes JA, Valero J, Cortes MJ, Labad A, Ochoa S, Ahuir M, Carlson J, Bernardo M, Canizares S, Escartin G, Canete J, Gallo P, Salamero M. Spanish adaptation of the Beck Cognitive Insight Scale (BCIS) for schizophrenia. Actas Esp Psiquiatr. 2012 Jan-Feb;40(1):2-9. Epub 2012 Jan 1. PMID 22344490
- [Background] Ochoa S, Lopez-Carrilero R, Barrigon ML, Pousa E, Barajas A, Lorente-Rovira E, Gonzalez-Higueras F, Grasa E, Ruiz-Delgado I, Cid J, Birules I, Esteban-Pinos I, Casanas R, Luengo A, Torres-Hernandez P, Corripio I, Montes-Gamez M, Beltran M, De Apraiz A, Dominguez-Sanchez L, Sanchez E, Llacer B, Pelaez T, Bogas JL, Moritz S; Spanish Metacognition Study Group. Randomized control trial to assess the efficacy of metacognitive training compared with a psycho-educational group in people with a recent-onset psychosis. Psychol Med. 2017 Jul;47(9):1573-1584. doi: 10.1017/S0033291716003421. Epub 2017 Feb 7. PMID 28166848
- [Background] Peralta V, Cuesta MJ. Psychometric properties of the positive and negative syndrome scale (PANSS) in schizophrenia. Psychiatry Res. 1994 Jul;53(1):31-40. doi: 10.1016/0165-1781(94)90093-0. PMID 7991730
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Wallwork RS, Fortgang R, Hashimoto R, Weinberger DR, Dickinson D. Searching for a consensus five-factor model of the Positive and Negative Syndrome Scale for schizophrenia. Schizophr Res. 2012 May;137(1-3):246-50. doi: 10.1016/j.schres.2012.01.031. Epub 2012 Feb 21. PMID 22356801
- [Background] Addington D, Addington J, Maticka-Tyndale E, Joyce J. Reliability and validity of a depression rating scale for schizophrenics. Schizophr Res. 1992 Mar;6(3):201-8. doi: 10.1016/0920-9964(92)90003-n. PMID 1571313
- [Background] Endicott J, Spitzer RL, Fleiss JL, Cohen J. The global assessment scale. A procedure for measuring overall severity of psychiatric disturbance. Arch Gen Psychiatry. 1976 Jun;33(6):766-71. doi: 10.1001/archpsyc.1976.01770060086012. PMID 938196
- [Background] World Health Organization (WHO). WHO Disability Assessment Schedule 2.0 (WHODAS 2.0). 2010 [Available from: http://www.who.int/classifications/icf/whodasii/en/]. Accessed 22 May 2019.
- [Background] Carlson J, Ochoa S, Haro JM, Escartin G, Ahuir M, Gutierrez-Zotes A, Salamero M, Valero J, Canizares S, Bernardo M, Canete J, Gallo P. Adaptation and validation of the quality-of-life scale: Satisfaction with Life Domains Scale by Baker and Intagliata. Compr Psychiatry. 2009 Jan-Feb;50(1):76-80. doi: 10.1016/j.comppsych.2008.05.008. Epub 2008 Aug 23. PMID 19059518
- [Background] Insel TR. Digital Phenotyping: Technology for a New Science of Behavior. JAMA. 2017 Oct 3;318(13):1215-1216. doi: 10.1001/jama.2017.11295. No abstract available. PMID 28973224
- [Background] Singh SP, Cooper JE, Fisher HL, Tarrant CJ, Lloyd T, Banjo J, Corfe S, Jones P. Determining the chronology and components of psychosis onset: The Nottingham Onset Schedule (NOS). Schizophr Res. 2005 Dec 1;80(1):117-30. doi: 10.1016/j.schres.2005.04.018. Epub 2005 Jun 22. PMID 15978778
- [Background] Cannon-Spoor HE, Potkin SG, Wyatt RJ. Measurement of premorbid adjustment in chronic schizophrenia. Schizophr Bull. 1982;8(3):470-84. doi: 10.1093/schbul/8.3.470. PMID 7134891
- [Background] Brett-Jones J, Garety P, Hemsley D. Measuring delusional experiences: a method and its application. Br J Clin Psychol. 1987 Nov;26(4):257-65. doi: 10.1111/j.2044-8260.1987.tb01359.x. PMID 3427248
- [Background] Corcoran R, Mercer G, Frith CD. Schizophrenia, symptomatology and social inference: investigating "theory of mind" in people with schizophrenia. Schizophr Res. 1995 Sep;17(1):5-13. doi: 10.1016/0920-9964(95)00024-g. PMID 8541250
- [Background] Gil D, Fernandez-Modamio M, Bengochea R, Arrieta M. [Adaptation of the Hinting Task theory of the mind test to Spanish]. Rev Psiquiatr Salud Ment. 2012 Apr-Jun;5(2):79-88. doi: 10.1016/j.rpsm.2011.11.004. Epub 2012 Jan 20. Spanish. PMID 22854578
- [Background] Baron-Cohen S, Wheelwright S, Jolliffe T. Is There a
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences. 2nd ed. New York: Routledge Academic; 1988.
- [Background] Cox D. Regression models and life tables (with discussions). J R Stat Soc. 1972;34:187-220.
- [Background] Lysaker PH, Roe D, Yanos PT. Toward understanding the insight paradox: internalized stigma moderates the association between insight and social functioning, hope, and self-esteem among people with schizophrenia spectrum disorders. Schizophr Bull. 2007 Jan;33(1):192-9. doi: 10.1093/schbul/sbl016. Epub 2006 Aug 7. PMID 16894025
- [Background] National Institute for Health and Clinical Excellence (NICE). Clinical Guidance 178 Schizophrenia and psychosis. 2014 [Available from: http://www.nice.org.uk/Guidance/CG178]. Accessed 22 May 2019.
- [Background] Drake RE, Gates C, Whitaker A, Cotton PG. Suicide among schizophrenics: a review. Compr Psychiatry. 1985 Jan-Feb;26(1):90-100. doi: 10.1016/0010-440x(85)90053-7. No abstract available. PMID 3881217
- [Background] Restifo K, Harkavy-Friedman JM, Shrout PE. Suicidal behavior in schizophrenia: a test of the demoralization hypothesis. J Nerv Ment Dis. 2009 Mar;197(3):147-53. doi: 10.1097/NMD.0b013e318199f452. PMID 19282679
- [Background] Schizophrenia Commission. The Abandoned Illness: A Report by the Schizophrenia Commission. Rethink Mental Illness, 2012.
- [Derived] Lopez-Morinigo JD, Barrigon ML, Porras-Segovia A, Ruiz-Ruano VG, Escribano Martinez AS, Escobedo-Aedo PJ, Sanchez Alonso S, Mata Iturralde L, Munoz Lorenzo L, Artes-Rodriguez A, David AS, Baca-Garcia E. Use of Ecological Momentary Assessment Through a Passive Smartphone-Based App (eB2) by Patients With Schizophrenia: Acceptability Study. J Med Internet Res. 2021 Jul 26;23(7):e26548. doi: 10.2196/26548. PMID 34309576
- [Derived] Lopez-Morinigo JD, Ruiz-Ruano VG, Martinez ASE, Estevez MLB, Mata-Iturralde L, Munoz-Lorenzo L, Sanchez-Alonso S, Artes-Rodriguez A, David AS, Baca-Garcia E. Study protocol of a randomised clinical trial testing whether metacognitive training can improve insight and clinical outcomes in schizophrenia. BMC Psychiatry. 2020 Jan 29;20(1):30. doi: 10.1186/s12888-020-2431-x. PMID 31996174